CLINICAL TRIAL: NCT02011256
Title: Early Detection Of Atrial Fibrillation In Patients With Transient Ischemic Attack - A Prospective Study
Brief Title: Early Detection Of Atrial Fibrillation In Patients With Transient Ischemic Attack
Acronym: NOTICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kenneth Pedersen, MD, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-20130027
Record Dates: First submitted 2013-12-09; First posted 2013-12-13 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Transient Ischemic Attack; Atrial Fibrillation
Keywords: Transient Ischemic Attack; Atrial Fibrillation; NOTICE; Implantable loop-recorder; Holter-monitoring
MeSH Terms: conditions — Ischemic Attack, Transient; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implantable loop-recorder (Experimental)
  Interventions: Device: Implantable loop-recorder

INTERVENTIONS:
Device: Implantable loop-recorder — All patients not diagnosed with atrial fibrillation with regular ECG or 72-hour Holter-monitoring will receive an ILR for 3 years.
  Other Names: Reveal XT, Medtronic Inc.

SUMMARY:
The purpose of this study is to determine the frequency of atrial fibrillation in patients with transient ischemic attack (TIA). Patients suffering TIA will have their heart rhythm extensively monitored with 72-hour Holter-monitoring and an implantable loop-recorder. Furthermore, the patients will be examined with echocardiography, coronary calcium-score and biomarkers with the purpose to predict which subjects at risk for developing atrial fibrillation.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and the survivors are often left with severe disability. Transient ischemic attack (TIA) is an episode of neurological dysfunction, but unlike stroke, the neurological deficits resolve completely within 24 hours. TIA and stroke share the same common underlying cause, and patients with a TIA are at high risk for developing a subsequent stroke. Atrial fibrillation (AF) is the most common cardiac arrhythmia and is recognized as the cause of around 25% of all strokes. The prevalence of AF rises with age, and it is estimated, that approximately 5-10% of all subjects over the age of 80 years has either persistent or paroxysmal AF. Regardless of the AF subtype the risk for stroke is the same, and oral anticoagulation therapy is recognized as a superior treatment of AF related stroke/TIA.

The goal of this project is to extend the normal workup of patients with TIA with a thorough heart monitoring program. This includes 72-hours ambulatory electrocardiogram and insertion of an implantable loop recorder (ILR). The ILR is small device implanted in the subcutaneous tissue in the left thoracic region. The device continuously monitors for arrhythmias in a period up to 3 years. The 150 patients enrolled will also receive an ultrasound examination of the heart and arteries of the neck and a computed tomography scan of the heart. Lastly, biomarkers with known or suspected association with stroke and AF will be measured.

The primary goal of the study is to determine, whether or not an extended heart monitoring program with an ILR will identify more patients with AF as the underlying cause of TIA. This can have enormous advantages for the patient, because the treatment with oral anticoagulation therapy reduces the risk of subsequent stroke by approximately 40% compared to conventional antiplatelet therapy. Secondly, the study means to identify patients at high risk for developing AF assessed with ultrasound, computed tomography and novel biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with TIA by a board certified neurologist
* Written consent
* Residents of Funen, Denmark or surrounding islands

Exclusion Criteria:

* Prior stroke
* Known atrial fibrillation
* Known contraindication for anticoagulant therapy
* Patients already in anticoagulant therapy
* Patients with estimated short life expectancy
* Pregnancy
* Prior TIA with known etiology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with TIA diagnosed with atrial fibrillation | 1 year
  All TIA-patients with no prior history of atrial fibrillation (AFLI) will be monitored for AFLI with 1) regular 12-lead ECG 2) 72-h Holter-monitoring and 3) implantable loop-recorder (ILR). If AFLI is diagnosed, then the patients will not receive further monitoring ie. not all patients will get Holter or ILR.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Pedersen, MD, Principal Investigator — University of Southern Denmark
Locations (1):
- Department of Cardiology, Odense Universityhospital, Odense, Funen, Denmark